CLINICAL TRIAL: NCT05411159
Title: The Effect of Opioid-free Anesthesia on PostOperative Nausea and Vomiting in Patients Undergoing Video-assisted Thoracoscopic Surgery: a Single-center Randomized Controlled Study
Brief Title: Effect of Opioid-free Anesthesia on PostOperative Nausea and Vomiting in Patients Undergoing Video-assisted Thoracoscopic Surgery
Acronym: OFA-PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Anshi Wu, Chief of department of Anesthesiology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022020817
Record Dates: First submitted 2022-05-30; First posted 2022-06-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Nausea and Vomiting; Opioid Use; Thoracic Diseases
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Thoracic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-Free Anesthesia (OFA froup) (Experimental): Opioid-free anesthesia group, avoid patients receive any kind of opioid during VATs.
  Interventions: Procedure: Opioid-Free Anesthesia (OFA)
- Standard general anesthesia (OA) (Active Comparator): Standard general anesthesia. Opioids allowed, including sufentanil, remifentanil, tramadol during VATs.
  Interventions: Procedure: Standard general anesthesia (OA)

INTERVENTIONS:
Procedure: Opioid-Free Anesthesia (OFA) — Opioid-free general anesthesia protocol:
  After entering the operating room, patients were given dexamethasone (5mg i.v.), atropine (0.25mg i.v.), flurbiprofen (50mg i.v.), dexmedetomidine (0.5ug/kg i.v. in 15min), and ultrasound-guided T4-5 paravertebral nerve block (0.5% Ropivacaine 20ml).
  Induction of anesthesia with lidocaine (1.5mg/kg i.v.), propofol (2-3mg/kg, i.v.), rocuronium (6-8mg i.v.).
  Intraoperative anesthesia was maintained by desflurane (0.5-1MAC), continuous intravenous infusion of dexmedetomidine (0.5ug/kg/h), and lidocaine (1.5mg/kg/h).
  Flurbiprofen (50 mg i.v.) given at the time of skin suture.
  Other Names: Non-Opioid anesthesia (NOA)
  Arms: Opioid-Free Anesthesia (OFA froup)
Procedure: Standard general anesthesia (OA) — Standard general anesthesia protocol:
  After entering the operating room, patients were given dexamethasone (5mg i.v.), atropine (0.25mg i.v.), flurbiprofen (50mg i.v.).
  Induction of anesthesia with lidocaine (1.5mg/kg i.v.), sufentanil (0.3-0.4ug/kg), propofol (2-3mg/kg, i.v.), rocuronium (6-8mg i.v. ).
  Intraoperative anesthesia was maintained by desflurane (0.5-1MAC) and continuous intravenous infusion of remifentanil (0.1-0.2ug/kg/min).
  Flurbiprofen (50 mg i.v.) given at the time of skin suture.
  Other Names: Opioid-based general anesthesia
  Arms: Standard general anesthesia (OA)

SUMMARY:
This study aimed to verify whether an Opioid-free Anesthesia (OFA) could effectively reduce the incidence of PONV after thoracoscopic-assisted surgery compared with standard general anesthesia (OA) regimens.

DETAILED DESCRIPTION:
Postoperative Nausea and Vomiting (PONV) is one of the most common complications after general anesthesia, which significantly reduces postoperative comfort and satisfaction of patients perioperatively. Meta-analysis showed that Opioid-free Anesthesia (OFA) significantly reduced the risk of postoperative PONV events in patients undergoing gynecology, breast, and abdominal surgery compared with standard general anesthesia (OA). The main hypothesis of the study is that an OFA could reduce the incidence of PONV in patients after thoracoscopic-assisted surgery than OA.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients planning elective thoracoscopic lobectomy or wedge resection under general anesthesia

Exclusion Criteria:

* ASA classification > 4
* BMI>35kg/m2
* Unable to communicate before surgery
* Received radiation therapy, chemotherapy, opioids or hormonal drugs within 14 days before surgery
* Anticipated intolerance to the anesthesia protocol of this study
* Expect prolonged mechanical ventilation after surgery
* Decline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 24 hours after surgery
  Assessed using Myles's simplified postoperative nausea and vomiting impact scale.
  The scale on the scale is a composite of the following 2 parts:
  (1) vomited or had dry-retching (0-3 points), and (2) nausea ( 0-3 points). (High scores represent severe).
  The score>0 is regarded as PONV occurred.

SECONDARY OUTCOMES:
The score of Simplified postoperative nausea and vomiting impact scale | 24 hours after surgery
  Assessed using Myles's simplified postoperative nausea and vomiting impact scale.
  The score on the scale is a composite of the following 2 parts:
  (1) vomited or had dry-retching score (0-3 points), and (2) nausea ( 0-3 points). (High scores represent severe)
Quality of post-operative recovery | 24 hours after surgery
  Assessed by the of quality of recovery-15 (QoR-15) scale. (0-150 points, High scores represent better)
Postoperative pain at rest and cough | 24 hours after surgery
  Assessed by the Numerical Assessment Scale (NRS) for pain. (0-10 points, High scores represent worse)
The six minute walking test (6MWT) | 48 hours after surgery
  Assessed by the 6MWT worksheet and report. (High scores represent better)

OTHER OUTCOMES:
Postoperative length of hospital stay | Up to 7 days after surgery
  Length of hospital stay in days
Postoperative anesthesia care unit (PACU) duration | Up to 4 hours after surgery
  PACU duration in minutes
Intraoperative complications | From entering to leaving the operating room, an average of 4 hours
  Assessed according to ClassIntra complication classifications
Postoperative Complications | within 7 days after surgery or discharge
  Assessed according to Clavien-Dindo surgical complication classifications
Health and well-being after surgery | 6 month after surgery
  Assessed according to the Short-Form (SF-36) health survey, included 36 items groups in 8 dimensions: physical functoning, physicial and emotional limitations, social functioning, bodily pain, general and mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The extent to which data is shared will be determined based on the progress of the study and local healthcare policies

REFERENCES:
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Dell-Kuster S, Gomes NV, Gawria L, Aghlmandi S, Aduse-Poku M, Bissett I, Blanc C, Brandt C, Ten Broek RB, Bruppacher HR, Clancy C, Delrio P, Espin E, Galanos-Demiris K, Gecim IE, Ghaffari S, Gie O, Goebel B, Hahnloser D, Herbst F, Ioannidis O, Joller S, Kang S, Martin R, Mayr J, Meier S, Murugesan J, Nally D, Ozcelik M, Pace U, Passeri M, Rabanser S, Ranter B, Rega D, Ridgway PF, Rosman C, Schmid R, Schumacher P, Solis-Pena A, Villarino L, Vrochides D, Engel A, O'Grady G, Loveday B, Steiner LA, Van Goor H, Bucher HC, Clavien PA, Kirchhoff P, Rosenthal R. Prospective validation of classification of intraoperative adverse events (ClassIntra): international, multicentre cohort study. BMJ. 2020 Aug 25;370:m2917. doi: 10.1136/bmj.m2917. PMID 32843333
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Derived] Yan X, Liang C, Jiang J, Ji Y, Wu AS, Wei CW. Effects of balanced opioid-free anesthesia on post-operative nausea and vomiting in patients undergoing video-assisted thoracic surgery: a randomized trial. BMC Anesthesiol. 2025 Feb 8;25(1):62. doi: 10.1186/s12871-025-02938-x. PMID 39923016
- [Derived] Yan X, Liang C, Jiang J, Ji Y, Wu A, Wei C. Effects of opioid-free anaesthesia on postoperative nausea and vomiting in patients undergoing video-assisted thoracoscopic surgery (OFA-PONV trial): study protocol for a randomised controlled trial. Trials. 2023 Dec 20;24(1):819. doi: 10.1186/s13063-023-07859-z. PMID 38124084